CLINICAL TRIAL: NCT03486015
Title: Oral Sweet Solution to Prevent Pain During Neonatal Hip Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 186081
Record Dates: First submitted 2018-02-07; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30% glucose (Experimental): This group will be given 2 ml of 30% glucose in the mouth before the physical examination of the infant.
  Interventions: Drug: 30% glucose
- Sterile water (Placebo Comparator): This group will be given 2 ml of sterile water in the mouth before the physical examination of the infant.
  Interventions: Drug: Sterile water

INTERVENTIONS:
Drug: Sterile water — 2 ml of sterile water
  Arms: Sterile water
Drug: 30% glucose — 2 ml of 30% glucose
  Arms: 30% glucose

SUMMARY:
This study evaluates the pain relieving effect of oral glucose during hip examinations on healthy, fullterm infants.

DETAILED DESCRIPTION:
All healthy, fullterm infants undergoes a medical examination after birth where 21 different components are assessed. One of the components is the hip examination which appears to be painful. Since painful experiences early in life can cause longterm negative effects it is important to treat pain during painful procedures.

One hundred healthy, fullterm infants were randomized to either glucose or sterile water orally before the routine medical examination before discharge from the maternity ward.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, fullterm infants that were undergoing a routine medical examination

Exclusion Criteria:

* Prematurity
* Parents inability to speak Swedish well enough to give consent
* Congenital malformations or other illnesses
* Any pain-relieving medicine administered in the previous 24 hours

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Pain will be measured with ALPS-Neo (Astrid Lindgren and Lund children's hospitals pain and stress assessment scale for preterm and sick newborn infants, range 0-10 where higher number means a higher intensity of rated pain) by a nurse | The assessment is made by the nurse when the physician starts with the hip examination, approximately 60 seconds after the study solution has been given.
  Pain assessment instrument
Pain will be measured by VAS (Visual analogue scale, range 0-10 where higher number means a higher intensity of rated pain) assessed by physician | The physician will make the VAS assessment directly after the physical examination is done, approximately 10 minutes after the study solution has been given.
  Pain assessment instrument
Pain will be measured by VAS (Visual analogue scale, range 0-10 where higher number means a higher intensity of rated pain) assessed by parent | The parents will make the VAS assessment directly after the physical examination is done, approximately 10 minutes after the study solution has been given.
  Pain assessment instrument
Total crying time will be measured | The total crying time is measured throughout the examination from zero minutes until approximately 10 minutes after the study solution has been given with the help of a stopwatch.
  Total amount of time (in minutes) the infant is crying during the examination.
Crying time during hip examination | The total crying time is measured from approximately 3 minutes from the study solution has been given until the hip examination has been completed (approx. during 30 sec up to 1 min) with the help of a stopwatch
  The amount of time (in minutes) the infant is crying during the hip examination.

IPD SHARING:
Plan to Share IPD: No